CLINICAL TRIAL: NCT03163810
Title: A Pilot Evaluation of the Effect of the Erchonia Verjú™ and EVRL Lasers on Reducing Aminoalanine Transaminase (ALT) in Individuals With Nonalcoholic Steatohepatitis (NASH)
Brief Title: A Study to See if Low Level Laser Light Therapy (LLLT) Can Improve the Condition of Nonalcoholic Steatohepatitis (NASH)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with recruitment
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC_NASH_PILOT
Record Dates: First submitted 2017-02-23; First posted 2017-05-23 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Erchonia Verju and EVRL Laser (Experimental): The Erchonia Verju Laser has 6 diodes that each emit 17 milliwatts (mW) 532 nanometers (nm) of green laser light.
  The Erchonia EVRL Laser emits 635 nanometers (nm) red light and 405 nm blue light simultaneously
  Interventions: Device: Erchonia Verju Laser; Device: Erchonia EVRL Laser

INTERVENTIONS:
Device: Erchonia Verju Laser — The Erchonia Verju Laser is applied 2 times a week to the front and back of the waist, hips and upper abdomen for 30 minutes each time over 8 to 12 weeks.
Device: Erchonia EVRL Laser — The Erchonia EVRL Laser is applied under the right ribcage angled towards the liver for 10 minutes, one time per week over the same 8 to 12 weeks as the Verju Laser is administered.

SUMMARY:
The purpose of this study is to determine whether low level laser therapy (LLLT) using the Erchonia VERJU and EVRL laser devices is effective in reducing aminoalanine transaminase (ALT) levels in individuals with nonalcoholic steatohepatitis (NASH).

DETAILED DESCRIPTION:
Nonalcoholic Fatty Liver Disease (NAFLD) is the most common liver disorder in the USA, present in 20% to 30% of the population and rapidly increasing. Fatty liver is generally diagnosed by abdominal ultrasound frequently as an incidental finding. Major risk factors for NAFLD include central (or abdominal) obesity, diabetes, elevated lipids, and metabolic syndrome.

Nonalcoholic steatohepatitis (NASH) are those patients where the presence of fat in the liver is accompanied by an inflammatory process that can cause progressive fibrosis in the liver. Which can ultimately lead to end stage liver disease (i.e., cirrhosis) and hepatic failure requiring liver transplantation. The 1990's was the decade of hepatitis C-related cirrhosis requiring transplantation. NASH is found in 3-5% of the population and is a subset of those patients with fatty liver.

Aminoaminoalanine Transaminase (ALT) is the liver enzyme measured in the blood that is a surrogate marker for inflammation and is frequently elevated in patients with NASH. Normalization of ALT is the ultimate treatment goal; however reduction in ALT is of significant clinical benefit.

Currently, the only treatment modality for patients with fatty liver disease is weight loss and exercise which is challenging for most patients. Therefore, a huge need exists for an alternative approach to reducing ALT levels for these patients.

Low level laser light therapy (LLLT) offers a simple, non-invasive, safe, effective and side-effect free alternative to achieving this goal, through LLLT's proven ability to effect weight loss, body circumference reduction and inflammation reduction.

Application of the Erchonia® Verjú™ (green diode) Laser and Erchonia 635nm (red light) lasers to the body mid-region has been proven through controlled clinical trials to reduce body circumference in these areas in a statistically significant and clinically meaningful manner and to effect a decrease in overall body weight, both associated with reducing in ALT levels for the management of NASH patients. The Erchonia® EVRL Laser violet diode has been proven in controlled clinical trials to additionally effect inflammation reduction, another factor important in the management of NASH patients. Additionally, the United States Food and Drug Administration (U.S. FDA) identifies the Erchonia 532nm (green diode) and 635nm (red diode) lasers under Product Code OLI as: "A Low Level Laser System for Aesthetic Use is a device using low level laser energy for the disruption of adipocyte cells within the fat layer for the release of fat and lipids from these cells for non-invasive aesthetic use."

Therefore, it is hypothesized that treatment application with the Erchonia LLLT devices will effect a reduction in body circumference, weight and inflammatory factors significant enough to effect a clinically meaningful decrease in ALT levels in NASH patients in a safe and timely manner.

The biochemical effect of Erchonia® low level laser light therapy devices stimulates the mitochondria of the adipocyte cells which in turn increases the production of adenosine triphosphate (ATP). The newly synthesized ATP triggers the up-regulation of cyclic adenosine monophosphate (cAMP). cAMP has been shown to stimulate cytoplasmic lipase, triggering the conversion of triglycerides into fatty acids and glycerol that can easily pass through the cell membrane. The transitory pore is evidence that the laser is allowing for the movement of fatty acids, glycerol, and triglycerides to pass across the membrane and into extra-cellular space. Through vasodilation of nearby blood vessels and arteries, oxidization of the triglycerides and fatty acids occurs within the extra-cellular space. Additionally, LLLT is known to influence the receptors on the membrane of the cell and on the membrane of the cell's mitochondrion, eventually reaching the cell's DNA, which directly controls cell function. When cells function better, so do tissues, and as such, LLLT promotes inflammation reduction and the consequent healing and regeneration of damaged tissues.

LLLT has been found to alter gene expression, cellular proliferation, intra-cellular (potential of hydrogen) phosphorus (pH) balance, mitochondrial membrane potential, generation of transient reactive oxygen species and calcium ion level, proton gradient and cellular oxygen consumption. With laser light able to induce cellular modulation, it has been proposed that LLLT may be able to serve as a subtle, non-invasive instrument in the reduction of clinical levels such as serum cholesterol levels, wherein it is proposed that laser therapy may suppress cholesterogenesis by altering the transcription factors responsible for the expression of essential genes involved in the biosynthetic process.

Recent studies have already identified the modulation of transcription factors subsequent to laser irradiation. Jackson and coworkers (2002) have identified more than twenty transcription factors that are regulated by the intracellular redox state. In a pilot study, Erchonia observed that low-level laser application 3 times per week for two weeks reduced cholesterol levels, and even more importantly, reduced LDL levels while preserving HDL levels. It is proposed that laser therapy, by means of altering the intracellular redox state, can affect the function of transcription factors tightly associated with cholesterol synthesis.

Moreover, laser therapy has been proven via multiple investigational studies to emulsify adipose tissue liberating all adipocyte stored fatty debris, demonstrated clinically through the observance of circumference reduction following LLLT administration. It is theorized that the liberation of fat is absorbed via the lymphatic system where lipolysis occurs in the lymph nodes and fatty-acid oxidation occurs in the liver. The mobilization of the fatty debris and production of ketone bodies may have an effect on applicable clinical lab markers.

Therefore, the Erchonia Lasers are proven to be efficacious in effecting weight loss, circumference reduction, reduction of inflammation and improvement in clinical levels, all of which are factors that both directly and indirectly impact the reduction of ALT levels and improvement in the overall condition of NASH in affected individuals.

ELIGIBILITY:
Inclusion Criteria:

* Review of subject's pre-existing medical records to confirm the current diagnosis of nonalcoholic steatohepatitis (NASH) according to the following criteria:

  * ALT elevated on two separate determinations
  * Abdominal ultrasound showing fatty liver
  * Blood work that excludes other potential etiologies of liver disease
* Subject has been on a stable diet and exercise regimen for NASH within the prior 6 months
* Subject agrees to maintain his or her current diet and exercise regimen throughout study participation
* Subject agrees to abstain from participating in any new treatments for NASH, other than the study treatments, throughout the course of study participation
* Elevated aminoalanine transaminase (ALT) level, defined as 20 or more Unites/Liter (U/L) above the normal gender-specific ALT levels: males: ALT ≥ 60 U/L; females: ALT ≥ 50 U/L

Exclusion Criteria:

* History of cardiovascular disease or events including, but not limited to, coronary artery disease, valvular heart disease, cardiac arrhythmias, congestive heart failure, myocardial infarction, stroke, transient ischemic attack, or peripheral vascular disease
* Cardiac surgeries or procedures, including but not limited to, coronary artery bypass surgery or stent placement, heart transplantation, pacemaker insertion or implantation of a defibrillator
* An implanted device in the target area to receive low level laser light therapy (e.g. pain pump, lap band, penile inflation device, ventriculo-peritoneal shunts, etc.)
* Known photosensitivity disorder
* Current active cancer or within one year of cancer treatment or remission
* Excessive alcohol consumption defined as 14 or more alcoholic drinks per week
* Pregnant, breastfeeding, or planning pregnancy prior to the end of study participation
* Serious mental health illness that in the opinion of the investigator would preclude the subject from study participation
* Active infection, wound or other external trauma to the target area to receive the laser therapy
* Developmental disability or cognitive impairment that in the opinion of the investigator would preclude adequate comprehension of the informed consent form and/or ability to record the necessary study measurements
* Involvement in litigation and/or a worker's compensation claim and/or receiving disability benefits related to NASH
* Participation in a clinical study or other type of research in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Percent (%) change from Baseline to Subject Study Endpoint evaluation in aminoalanine transaminase (ALT) level. | 2 or 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Schron, MD, Principal Investigator
Locations (1):
- Meridian Integrative Medicine, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No